CLINICAL TRIAL: NCT03300076
Title: Multicenter, Open-label, Non Interventional, Prospective, Observational Clinical Trial to Assess the Compliance and Quality of Life in Greek Asthmatic Patients
Brief Title: COMPLliancE and qualiTy of lifE in Asthma
Acronym: COMPLETE
Status: Completed | Type: Observational
Sponsor: Elpen Pharmaceutical Co. Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 2017-HAL-EL-74
Record Dates: First submitted 2017-09-28; First posted 2017-10-03 (Actual); Last update posted 2018-12-05 (Actual); Status verified 2018-03

CONDITIONS: Asthma; Compliance, Patient; Quality of Life
MeSH Terms: conditions — Asthma; Patient Compliance

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A multicenter, open, non-interventional, prospective, clinical observational study on Conformity to Therapy and Quality of Life in Asthma in patients living in Greece

DETAILED DESCRIPTION:
Dry powder devices, available since 1970, have been developed to make inhalation simpler than pMDIs and relieve the need for co-ordination of spraying and inhalation, which is particularly important for patient groups such as the elderly and children. In addition, dry powder devices do not contain propellant gases potentially hostile to the environment as they are activated by inhalation of the patient and do not cause cold sensation upon inhalation.

Today, the combination of inhaled corticosteroid (ICS) and long-acting β2-inducer with an inhaler is the basic treatment for asthma6.

The addition of long-acting β2-inducer (LABA) to a daily inhaled corticosteroid regimen1:

* Improves the symptoms,
* Reduces nightly asthma symptoms,
* Improves pulmonary function,
* Reduces the use of β2-agonists for rapid action,
* Reduces the number of seizures,
* Does not increase the risk of hospitalizations due to asthma,
* Achieves clinical asthma control in more patients, faster and with less ICS than would be required if ICS were administered alone.

The greater effectiveness of combination therapy has led to the development of stable combination inhalers that both glucocorticosteroids and LABA (eg, fluticasone-salmeterol, budesonide-formoterol stable compounds) are concomitantly conveyed.

Stable combinations are more user-friendly for patients, potentially increasing compliance, and ensure that LABA is always accompanied by glucocorticosteroid1. Of the combinations available, the budesonide-formoterol combination can be used both as maintenance therapy and symptom relief due to the rapid onset of formoterol compared to salmeterol. Both components of the budesonide-formoterol combination when administered are helpful in enhancing protection from severe seizures in patients receiving combination therapy for maintenance and improve the control of asthma at relatively low ICS doses.

ELIGIBILITY:
Inclusion Criteria:

* Male or female asthma patients over 18 years of age
* Compliance with treatment
* Compliance with study procedures
* Signed informed consent form
* Patients not satisfactorily controlled with inhaled corticosteroids and the use of inhaled short-acting β2-primers or patients already adequately controlled with both inhaled corticosteroids and long-acting β2-stimulants:

  1. Patients receiving ICS inhaled and SABA invoked
  2. Patients receiving inhaled ICS and LABA with separate devices each
  3. Patients receiving periodic and not continuously stable combination of ICS and LABA but not being treated for at least 1 month
  4. Patients who did not receive any treatment and the doctor decides to immediately start the fixed combination of ICS and LABA

Exclusion Criteria:

* Male or female asthma patients under 18 years of age
* Unsigned patient consent
* Non-compliance with treatment
* Non-compliance in study procedures
* COPD patients (at any stage)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Asthmatic adult patients
Sampling Method: Non-Probability Sample
Enrollment: 800 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
Quality of Life | 6 months
  Change in mini AQLQ scale

SECONDARY OUTCOMES:
Compliance | 6 months
  Change in MMAS-8 scale

CONTACTS AND LOCATIONS:
Locations (1):
- Sotiria Pulmonary Hospital, Athens, Greece

REFERENCES:
- [Derived] Exarchos KP, Rovina N, Krommidas G, Latsios D, Gogali A, Kostikas K. Adherence and quality of life assessment in patients with asthma treatment with budesonide/formoterol via the Elpenhaler device: the COMPLETE study. BMC Pulm Med. 2022 Jun 27;22(1):254. doi: 10.1186/s12890-022-02049-0. PMID 35761234